CLINICAL TRIAL: NCT05844917
Title: Ultrasound-Based Detection Of Subclinical Arthritis Among Patients With Systemic Lupus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aya Abdelsabor Abdelbaset, Sohag Egypt, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: U/S arthritis in SLE
Record Dates: First submitted 2023-04-16; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Ultrasound
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 50 character (Experimental)
  Interventions: Device: ultrasound

INTERVENTIONS:
Device: ultrasound — Ultrasound detection of subclinical arthritis among Patients With SLE

SUMMARY:
The aim of this study is to assess the prevalence and precise grading of US abnormalities of the hand and wrist in asymptomatic patients with SLE, while comparing these findings with a group of patients with SLE with musculoskeletal signs or symptoms and with healthy controls.

DETAILED DESCRIPTION:
Systemic Lupus Erythematosus (SLE) is a chronic inflammatory autoimmune disorder associated with a wide range of symptoms and physical findings. It is characterized by loss of tolerance to self-antigens, formation of immune complexes, and an activated type I interferon system .

Joint involvement is one of the most common features of systemic lupus erythematosus (SLE), with up to 95% of patients experiencing arthralgia or arthritis during the course of their disease .

While multiple joints can be affected, nearly 50% of patients report difficulties in daily life performance due to hand symptoms .

Traditionally, SLE arthritis is considered to be mild, reversible and non-erosive, with only 5-15% of cases progressing to deforming arthropathy, either erosive-as in rhupus syndrome (an overlap of SLE with rheumatoid arthritis (RA))-or non-erosive-as in Jaccoud's arthropathy .

In routine clinical practice, joint involvement is usually assessed with physical examination and radiographical studies. However, this approach has been shown to have a low sensitivity for joint abnormalities when compared with ultrasound (US) evaluation or MRI, suggesting that the burden of joint inflammation may be underestimated in the current clinical practice .

The value of US with power Doppler (PD) in inflammatory arthritis has been extensively demonstrated in the literature, with similar sensitivity and specificity in the detection of synovitis in comparison with MRI, with the advantage of being more accessible and less expensive .

While US shows the morphology of the synovial membrane, PD identifies increased vascularisation within it, allowing for the detection of active joint inflammation. It is known that in RA synovial abnormalities are present before clinically evident arthritis develops, and that early treatment can limit erosive changes and avoid disease progression. In this context, US PD has nowadays an established role in the detection of subclinical joint inflammation in RA, namely to predict progression in patients with clinical remission .

Although there is evidence that US PD is a valuable technique in the evaluation of musculoskeletal symptoms in SLE, the prevalence of subclinical joint abnormalities in SLE remains to be defined.

Furthermore, while it is known that minimal synovial proliferation may be seen in up to 50% of healthy subjects, the distinction between 'normal' synovial hypertrophy (SH) and pathological subclinical synovitis in SLE still requires clarification .

ELIGIBILITY:
Inclusion Criteria:

* Cases diagnosed as SLE according to the 2019 ACR/EULAR classification criteria.
* Agreeing to be included in the study
* Age >18 years

Exclusion Criteria:

* Patients with clinical SLE arthritis
* Patients of Rhupus and patients with any collagen disease that causes arthritis other than systemic lupus erythematosus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
subclinical arthritis | 6 months
  detection of subclinical arthritis by ultrasound in SLE patients

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

REFERENCES:
- [Background] Aringer M, Costenbader K, Daikh D, Brinks R, Mosca M, Ramsey-Goldman R, Smolen JS, Wofsy D, Boumpas DT, Kamen DL, Jayne D, Cervera R, Costedoat-Chalumeau N, Diamond B, Gladman DD, Hahn B, Hiepe F, Jacobsen S, Khanna D, Lerstrom K, Massarotti E, McCune J, Ruiz-Irastorza G, Sanchez-Guerrero J, Schneider M, Urowitz M, Bertsias G, Hoyer BF, Leuchten N, Tani C, Tedeschi SK, Touma Z, Schmajuk G, Anic B, Assan F, Chan TM, Clarke AE, Crow MK, Czirjak L, Doria A, Graninger W, Halda-Kiss B, Hasni S, Izmirly PM, Jung M, Kumanovics G, Mariette X, Padjen I, Pego-Reigosa JM, Romero-Diaz J, Rua-Figueroa Fernandez I, Seror R, Stummvoll GH, Tanaka Y, Tektonidou MG, Vasconcelos C, Vital EM, Wallace DJ, Yavuz S, Meroni PL, Fritzler MJ, Naden R, Dorner T, Johnson SR. 2019 European League Against Rheumatism/American College of Rheumatology Classification Criteria for Systemic Lupus Erythematosus. Arthritis Rheumatol. 2019 Sep;71(9):1400-1412. doi: 10.1002/art.40930. Epub 2019 Aug 6. PMID 31385462
- [Background] Aringer M, Costenbader K, Daikh D, Brinks R, Mosca M, Ramsey-Goldman R, Smolen JS, Wofsy D, Boumpas DT, Kamen DL, Jayne D, Cervera R, Costedoat-Chalumeau N, Diamond B, Gladman DD, Hahn B, Hiepe F, Jacobsen S, Khanna D, Lerstrom K, Massarotti E, McCune J, Ruiz-Irastorza G, Sanchez-Guerrero J, Schneider M, Urowitz M, Bertsias G, Hoyer BF, Leuchten N, Tani C, Tedeschi SK, Touma Z, Schmajuk G, Anic B, Assan F, Chan TM, Clarke AE, Crow MK, Czirjak L, Doria A, Graninger W, Halda-Kiss B, Hasni S, Izmirly PM, Jung M, Kumanovics G, Mariette X, Padjen I, Pego-Reigosa JM, Romero-Diaz J, Rua-Figueroa Fernandez I, Seror R, Stummvoll GH, Tanaka Y, Tektonidou MG, Vasconcelos C, Vital EM, Wallace DJ, Yavuz S, Meroni PL, Fritzler MJ, Naden R, Dorner T, Johnson SR. 2019 European League Against Rheumatism/American College of Rheumatology classification criteria for systemic lupus erythematosus. Ann Rheum Dis. 2019 Sep;78(9):1151-1159. doi: 10.1136/annrheumdis-2018-214819. Epub 2019 Aug 5. PMID 31383717
- [Background] Ball EM, Bell AL. Lupus arthritis--do we have a clinically useful classification? Rheumatology (Oxford). 2012 May;51(5):771-9. doi: 10.1093/rheumatology/ker381. Epub 2011 Dec 15. PMID 22179731
- [Background] Bresnihan B, Kane D. Sonography and subclinical synovitis. Ann Rheum Dis. 2004 Apr;63(4):333-4. doi: 10.1136/ard.2003.015982. No abstract available. PMID 15020323